CLINICAL TRIAL: NCT05973266
Title: The Effect of Mobile Application-Based Bowel Preparation Training on the Patient's Bowel Preparation Compliance, Quality and Anxiety Level in Patients for Whom Colonoscopy is Planned
Brief Title: The Effect of Mobile Application-Based Bowel Preparation Training on the Patient's Education Whom Colonoscopy is Planned
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kubra Sengor (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor-Investigator, Kubra Sengor, Research Assistant, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: IstanbulUC-FNHF-KS-01
Record Dates: First submitted 2023-07-26; First posted 2023-08-02 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Colon Disease; Colon Cancer
Keywords: colonoscopy; bowel preparation; mobile application
MeSH Terms: conditions — Colonic Diseases; Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental design
Who Masked: Outcomes Assessor
Masking Description: endoscopist blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Patients using mobile application as well as verbal and written information in bowel preparation training in patients who will undergo colonoscopy will constitute the experimental group.
  Interventions: Behavioral: Mobile Application-Based Bowel Preparation Training
- Control Group (No Intervention): Patients who will be given oral and written information in bowel preparation training in patients who will undergo colonoscopy will form the control group.

INTERVENTIONS:
Behavioral: Mobile Application-Based Bowel Preparation Training — The contents of the training in the mobile application where the patients receive bowel preparation training before the procedure are; short videos, images and slides about colonoscopy, bowel preparation drugs, liquid-clear diet and foods recommendations.A mobile application-based training will be provided to guide patients, where user (patient) usage activities are monitored by the researcher, sending notifications or reminders to the patient in accordance with the colonoscopy procedure date.
  Arms: Experimental Group

SUMMARY:
Colonoscopy is the examination of the large intestine with an instrument called a colonoscope. To make an accurate evaluation during a colonoscopy performed for diagnosis and treatment, adequate preparation of the large intestine must be made. Information given to patients is very important for adequate bowel preparation and adherence to treatment.

Therefore, this study was planned as a prospective, single-blind randomized controlled study to determine the effect of mobile application-based bowel preparation training on patients' bowel preparation compliance, quality and anxiety level in patients scheduled for colonoscopy.

The study will be carried out with 160 patients (experimental: 80, control: 80) who will apply to the Istanbul University Istanbul Medical Faculty Hospital General Surgery Department Endoscopy Unit, who will undergo colonoscopy as an outpatient.

Both groups will receive oral and written instructions for bowel preparation. In addition, the smart phone app group will received instructions through a medical smart phone app. The primary outcome was the rate of adequate bowel preparation according to the Boston bowel preparation scale score. The secondary outcomes included patient compliance.

DETAILED DESCRIPTION:
Colorectal cancers (CRC) are the third most common cancers worldwide, regardless of age and gender, and the second among cancer deaths. In terms of the incidence of colorectal cancers in Turkey, regardless of gender, it ranks third in all age groups (9.8% in men, 8.1% in women) (Turkey Unified Database, 2017). According to the Global Cancer 2020 data published by the International Agency for Research on Cancer (IARC), it is predicted that approximately 21,000 individuals will be diagnosed with colorectal cancer in 2020 and the estimated age-standardized death rate will be 10.1 per 100,000 individuals. Colonoscopy, which is the gold standard for early diagnosis of colorectal cancers, reduces cancer-related morbidity and mortality rates (World Health Organization, 2022).

Colonoscopy is a lower gastrointestinal system endoscopy method that enables imaging of the large intestine (colon) for the purposes of screening, diagnosis, treatment and monitoring of colorectal and anal canal pathologies. In the colonoscopy procedure, adequate intestinal preparation is necessary for a good visualization of the entire mucosa and for an accurate evaluation. American Society for Gastrointestinal Endoscopy (ASGE), ideal bowel preparation (BH); defined as the rapid clearance of all macroscopic and microscopic fecal load in the colon without disturbing the patient's comfort and fluid-electrolyte balance.

Inadequate bowel cleansing rates ranging from 10% to 75% have been reported in studies. It is stated that when the bowel preparation of the patients is insufficient, 45% less polyps are detected, and the rate of incomplete and canceled procedures is 5%. In addition, gas compression and explosion, which can be seen rarely as a result of gas insufflation during colonoscopy due to insufficient bowel preparation, can cause perforation of the intestines and undesirable events such as bleeding. As a result, inadequate bowel cleansing can cause repetition or prolongation of the procedure, loss of labor, time and cost for patients and healthcare personnel.

Before colonoscopy, nurses provide patients with written and oral bowel preparation standard training set by the institution. However, many studies suggest that this training should be supported by visual and auditory tools to increase its effectiveness. In interventional studies aimed at increasing the effectiveness of colonoscopy bowel preparation, the use of educational booklets, patient education with poster images, patient education with both visual use and educational videos, telephone/short message, interactive social media and patient education with the use of telephone applications methods were used.

As a result of the literature review, Mobile Application Based Bowel Preparation Training, which is an innovative method, was planned in order to improve the quality of colonoscopy bowel preparation. In this study, it was determined that the quality of bowel preparation and compliance with the procedure will increase by applying Mobile Application-Based Bowel Preparation Training together with the standard education method in patient education before colonoscopy; anxiety is predicted to decrease.

Aim This study was planned as a prospective, single-blind randomized controlled study to determine the effect of mobile application-based bowel preparation training on patients' bowel preparation compliance, quality and anxiety level in patients scheduled for colonoscopy. With the increase in the quality of bowel preparation, effective and accurate evaluation of colon pathologies during colonoscopy and, as a result, early diagnosis of colon cancer will be provided. With adequate bowel preparation, the risk of complications (perforation, hemorrhage, etc.) that may occur during colonoscopy will be reduced, and labor, time and cost loss due to repeated or prolonged colonoscopy will be prevented.

Material Method In this study, in order to determine the effect of mobile application-based bowel preparation training on the quality of bowel preparation, compliance and anxiety level of patients who are planned for colonoscopy; The calculation (d-value) method developed by Cohen was used to calculate the effect size. To determine the effect size index d. The findings of the study, which investigated the effect of mobile application on patient bowel cleansing before colonoscopy, were used. In the calculation made using the findings of this study, the effect size of the bowel cleansing efficiency between the two groups (Experiment=7.70±1.1; Control=7.70±0.8; p=0.007) was determined to be d=0.48. In this context, a sample group of 140 people, 70 people in each group, was determined with the help of the G-power (version 3.1) package program, accompanied by the specified criteria, with d=0.48, α=0.05 (error margin), 1-β=0.80 (power). Due to the loss of patients who left the study during data collection, 10 individuals will be added to the experimental and control groups, and the data collection process will be completed. The sample will consist of patients who meet the inclusion criteria and agree to participate in the study, whose colonoscopy procedure is planned.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years to 65 Years, Internet-enabled smart phone Outpatient admission to endoscopy Patient undergoing colonoscopy for the first time Patients who agreed to participate in the study

Exclusion Criteria:

* Have undergone colon and abdominal surgery Active lower gastrointestinal bleeding Known dementia etc. patients with cognitive disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-06-03 (Actual); Primary Completion 2023-10-27 (Estimated); Study Completion 2023-12-29 (Estimated)

PRIMARY OUTCOMES:
quality of bowel preparation | filled in by the endoscopist during the colonoscopy procedure after training
  The Boston bowel preparation scale is a four-point (0-3) assessment tool for bowel cleansing administered separately for each of the three sections of the colon during colonoscopy.Each region of the colon receives a "segment score" from 0 to 3 and these segment scores are summed for a total Boston bowel preparation scale score ranging from 0 to 9. Therefore, the maximum Boston bowel preparation scale score for a perfectly clean colon without any residual liquid is 9 and the minimum Boston bowel preparation scale score for an unprepared colon is 0.

SECONDARY OUTCOMES:
Anxiety | will be administered to patients before colonoscopy
  State-Trait Anxiety Inventory (STAI); STAI-I was developed by Spielberger in 1970. The scale consists of 20 items. The answers range from 1-4. The total point value obtained from the scale is between 20-80. A high score indicates a high level of anxiety. STAI 2 Trait Anxiety Scale; It aims to measure how the individual feels, that is, his trait anxiety, regardless of the situation and conditions he is in. These individuals also experience state anxiety more frequently and intensely than others. In answering the state anxiety scale; choosing one of the options "Not at all", "A little", "A lot", "Totally" according to the level of severity of the feelings, behaviors or thoughts expressed by the items; In answering the trait anxiety scale, it is required to select and mark one of the options "Almost Never", "Sometimes", "Very Often" and "Almost Always" according to the frequency level of the feelings, behaviors or thoughts expressed by the items.

CONTACTS AND LOCATIONS:
Overall Officials: Kübra Şengör, Msc, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University - Cerrahpasa (IUC), Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Sengor K, Keskin M, Akyuz N. Mobile app-based bowel preparation training: effects on compliance, quality, and anxiety in colonoscopy patients-a randomized controlled trial. Surg Endosc. 2025 Nov;39(11):7312-7323. doi: 10.1007/s00464-025-12074-9. Epub 2025 Aug 27. PMID 40866593